CLINICAL TRIAL: NCT04225286
Title: Intranasal Human Milk as Stem Cell Therapy in Preterm Infants With Intraventricular Hemorrhage
Brief Title: Intranasal Human Milk for Intraventricular Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Principal Investigator, Rebecca Hoban, MD MPH, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1911
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Intraventricular Hemorrhage
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal human breast milk (Experimental): Human breast milk delivered intranasally to preterm infants (<33 weeks gestation at birth, stratified < and ≥28 weeks) with any grade IVH/intraparenchymal hemorrhage/infarction identified on head ultrasound in the first 10 days of life.
  Dosing: Escalating dose starting at 0.2mL into one nostril with repeat dose 10-15 minutes later 1-2x daily, depending on availability of fresh HM
  Interventions: Other: Human breast milk

INTERVENTIONS:
Other: Human breast milk — Intranasal human breast milk

SUMMARY:
Intraventricular hemorrhage (IVH) is a leading cause of brain injury in infants born before term. Severe IVH, which occurs nearly exclusively in very preterm infants (born before 32 weeks gestation) who are already at risk of neurodevelopmental delays and cerebral palsy at baseline, results in a ~5 times higher risk of death or moderate-severe neurodevelopmental impairment, as well as short-term morbidities in the neonatal intensive care unit (NICU). Infants with grade I and II IVH, although less severe than the higher grades of IVH, also have a higher risk of death or moderate to severe neurodevelopmental impairment compared to infants with a normal head ultrasound. Outcomes are worsened by the fact that the brains of these preterm infants are not fully developed, so the progenitor cells that would later differentiate and mature are damaged, resulting in hypomyelination and gray matter loss that are associated with poor neurodevelopmental outcomes. There is no available therapy to treat the IVH or resultant brain injury, other than symptomatic management for resultant post-hemorrhagic hydrocephalus with lumbar punctures and temporary or permanent shunts, which have significant risks on their own.

This is a phase I trial to determine whether fresh intranasal human milk (HM) can be safely delivered as stem cell therapy to preterm IVH patients within a 3-hour window from HM expression and to identify signals which would indicate whether intranasal HM stimulates the repair of damaged brain tissue. Outcomes will be compared to HM fed historical IVH controls. Recruitment will take place in tertiary care NICUs in Toronto, which care for the highest proportion of very preterm infants with IVH in Canada. These NICUs have already adopted a common protocolized approach to manage severe IVH and post-hemorrhagic hydrocephalus with intensive monitoring, early symptomatic management, and detailed prospectively collected IVH data.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants (<33 weeks gestation at birth, stratified < and ≥28 weeks) with any grade IVH/intraparenchymal hemorrhage/infarction on head ultrasound in the first 10 days of life. Diagnostic criteria will be based on the Papile definitions as used by the study sites/Toronto Centre for Neonatal Health for PHVD management, outlined in the document "Intraventricular Hemorrhage and Measurements of Lateral Ventricular Size from Head Ultrasound"

Exclusion Criteria:

1. Disorders associated with neurodevelopmental delays or impairment (i.e. Trisomy 21)
2. Moribund/critically ill infant or known lethal diagnosis with plans by medical team to redirect care
3. Choanal atresia or anomalies that would not allow intranasal treatment
4. Surgical condition (e.g. esophageal atresia) for which team feels intranasal HM is contraindicated
5. Enrolled in other intervention trials in which primary target is neurodevelopmental outcome
6. Parent with lactation contraindication(s) (i.e. HIV) or parent who declines lactation initiation
7. Lactating parent unable to provide fresh HM: unable/unwilling to pump at study site or unable to have fresh HM delivered by designee at least once/day for 3 days within 3 hours of pumping AND located (in hospital or home) >30km from study sites (for courier services)

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as described in the protocol | 1 year
  Increased respiratory support settings or increase in Fio2 by more than 10% for more than 1 hour after the intervention, need for PPV/bagging immediately (within 5 minutes) of administration, or need for escalation of respiratory modality (ie NC to CPAP or NIV to intubation) in the hour after administration.

SECONDARY OUTCOMES:
The number of participants with IVH related long-term adverse neurodevelopmental outcomes compared with a cohort of HM-fed historical controls with IVH from 30 months prior to the intervention cohort. | 2 years
  Cerebral Palsy, Gross motor delay (in the absence of CP), Fine motor delay, Vision impairment (blindness or wears glasses), Hearing impairment (aided / cochlear implant), Cognitive delay, Speech and language delay
Interference of IHM administration with routine clinical care measured using post-intervention staff survey | 1 year
Number of participants with any grade IVH unable to be recruited within 10 days of birth | 1 year
Number of eligible patients unable to receive intranasal HM administration within 3 hours of HM collection | 1 year

OTHER OUTCOMES:
Number of stem cells in maternal milk provided by lactating parents of preterm infants | 1 year
Number of stem cells measured in CSF of treated infants who have lumbar punctures for clinical indications. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Hoban, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Gallipoli A, Unger S, El Shahed A, Fan CS, Signorile M, Wilson D, Hoban R. Outcomes after intranasal human milk therapy in preterm infants with intraventricular hemorrhage. J Perinatol. 2025 Feb;45(2):202-207. doi: 10.1038/s41372-024-02147-3. Epub 2024 Oct 9. PMID 39384614
- [Derived] Hoban R, Gallipoli A, Signorile M, Mander P, Gauthier-Fisher A, Librach C, Wilson D, Unger S. Feasibility of intranasal human milk as stem cell therapy in preterm infants with intraventricular hemorrhage. J Perinatol. 2024 Nov;44(11):1652-1657. doi: 10.1038/s41372-024-01982-8. Epub 2024 Apr 30. PMID 38688998